CLINICAL TRIAL: NCT01239316
Title: A Phase II Clinical Trial Evaluating the Efficacy and Safety of GDC-0449 in Children With Recurrent or Refractory Medulloblastoma
Brief Title: Vismodegib in Treating Younger Patients With Recurrent or Refractory Medulloblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02546; NCI-2011-02546 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000688451; PBTC-032; PBTC-032 (Other: Pediatric Brain Tumor Consortium); PBTC-032 (Other: CTEP); U01CA081457 (NIH)
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-04

CONDITIONS: Recurrent Childhood Medulloblastoma
MeSH Terms: conditions — Medulloblastoma | interventions — HhAntag691

ARMS (1):
- Treatment (vismodegib) (Experimental): Patients receive vismodegib PO QD on days 1-28. Treatment repeats every 28 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Vismodegib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC-0449; Hedgehog Antagonist GDC-0449

SUMMARY:
This phase II trial studies how well vismodegib works in treating younger patients with recurrent or refractory medulloblastoma. Vismodegib may slow the growth of tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the efficacy of GDC-0449 (vismodegib) treatment for pediatric patients with recurrent or refractory medulloblastoma, as measured by the sustained objective response rates for patients without (stratum A) and with (stratum B) evidence of activation of Hedgehog (Hh) signaling pathway in their tumors.

II. Characterize the pharmacokinetics (plasma) of GDC-0449 in children/adolescents with refractory medulloblastoma.

III. To document pathologic and genomic methods to identify medulloblastomas with activation of the Hh signaling pathway.

SECONDARY OBJECTIVES:

I. Document and describe toxicities associated with GDC-0449 administered on a daily schedule.

II. Estimate the duration of objective response and progression-free survival (PFS).

III. Characterize the pharmacokinetics (cerebrospinal fluid) of GDC-0449 in children/adolescents with refractory medulloblastoma.

OUTLINE: This is a multicenter study. Patients are stratified according to evidence of activation of Hedgehog signaling pathway in their tumors (without vs with vs unknown).

Patients receive vismodegib orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.

Plasma and cerebrospinal fluid samples are collected periodically for pharmacokinetic and other correlative studies.

After completion of study treatment, patients are followed up every other month for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed diagnosis of medulloblastoma that is recurrent, progressive, or refractory to standard therapy and for which there is no known curative therapy
* Patient must have adequate archival formalin fixed, paraffin embedded (FFPE) primary tumor material for biology studies; specifically, adequate archival FFPE tumor material is either:

  * An FFPE block, preferably in which tumor occupies an area of at least 10x10 mm if available, and is free of surgical or processing artifacts; tumor in the submitted FFPE block must not have been obtained from the CUSA trap OR
  * Preferably15x5µm sections if available from an FFPE tissue block conforming to the above criteria AND
  * Tissue submission must be accompanied by a copy of the pathology report
* Patients must have bi-dimensionally measureable disease in the brain or spinal cord defined as at least one lesion that can be accurately measured in at least 2 planes in order to be eligible for this study
* Patients must have a body surface area (BSA) of >= 0.67m^2 and at most 2.5m^2
* Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration; this is to be documented in the database
* Karnofsky performance status of >= 50% in patients > 16 years, or Lansky performance status of >= 50% in patients >= 3 yrs and =< 16 years, assessed within two weeks prior to registration
* Must have recovered from prior treatment-related toxicity; no other myelosuppressive chemotherapy or immunotherapy within 4 weeks prior to study entry (6 weeks if prior nitrosurea)
* Decadron dose should also be stable or decreasing for at least 1 week (7days) prior to starting therapy
* Radiation therapy (XRT) >= 3 months prior to study entry for craniospinal irradiation; >= 8 weeks for local irradiation to primary tumor; >= 2 weeks prior to study entry for focal irradiation for symptomatic metastatic sites
* Off all colony stimulating factors > 1 week prior to study entry (granulocyte colony stimulating factor [GCSF], granulocyte macrophage colony stimulating factor [GM CSF], erythropoietin)
* Prior therapy will include primary therapy (including radiation therapy and chemotherapy) and a maximum of 2 additional salvage therapies; patients can enroll on the protocol after failure on primary therapy
* Absolute neutrophil count (ANC) >= 1000 µL
* Platelet count >= 50,000/uL (transfusion independent)
* Hemoglobin >= 8.0 gm/dL (may receive red blood cell [RBC] transfusions)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70ml/min/1.73 m^2 or a serum creatinine =< 1.5 mg/dL
* Serum Total Bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 times institutional ULN for age
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2.5 times institutional ULN for age
* Alkaline Phosphatase =< 1.5 times institutional ULN
* Serum albumin >= 2.5 g/dL
* Patient must have recovered from the significant acute toxicities of all prior therapy before entering this study and meet all other eligibility criteria specified in the Inclusion and Exclusion Criteria
* Pregnancy should be avoided for 12 months after the last dose of GDC-0449 for females of child-bearing potential; female patients of childbearing potential must not be pregnant or breast-feeding; female patients of childbearing potential must have a negative serum or urine pregnancy test within 24 hours prior to beginning treatment
* Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 10-14 days and within 24 hours prior to the first dose of GDC-0449 (serum or urine); a pregnancy test (serum or urine) will be administered every 4 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of GDC-0449; prior to dispensing GDC-0449, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the of GDC-0449 to cause spontaneous abortion or birth defects; female patients are required to use two forms of acceptable contraception, including one barrier method during participation in the study and for the 12 months following the last dose; all patients should receive contraceptive counseling either by the investigator, or by an obstetrician (OB), gynecologist or other physician who is qualified in this area of expertise; if a woman of childbearing potential believes that her contraceptive method has failed, emergency contraception should be considered; if a patient is suspected to be pregnant, GDC-0449 should be immediately discontinued; in addition, a positive urine test must be confirmed by a serum pregnancy test; if it is confirmed that the patients is not pregnant, the patient may resume dosing with GDC-0449; if a female patient becomes pregnant during therapy or within 12 months after the last dose of GDC-0449, or if the female partner of a male patient exposed to the drug becomes pregnant while the male patient is receiving GDC-0449 or within 12 months after the last dose of GDC-0449, the investigator must be notified in order to facilitate outcome follow-up; female patients should not breastfeed a baby while on this study; female patients must NEVER donate ova while being treated with GDC-0449; all sexually active male subjects (including those who have undergone vasectomy) should utilize a barrier form of contraception during study treatment and for 12 months after the last dose as it is not known whether GDC-0449 that may be present in seminal fluid would cause serious or life-threatening birth defects in a fetus born to the female partner of a male subject; males should also not donate sperm during treatment or up to 12 months after the last dose
* Signed informed consent must be obtained including for pharmacokinetic study according to institutional guidelines

Exclusion Criteria:

* Central nervous system (CNS) embryonal tumor other than medulloblastoma; for example, patients with diagnosis of Atypical Teratoid / Rhabdoid Tumor (ATRT), primitive neuroectodermal tumor (PNET) from a non-cerebellar site within the central nervous system, ependymoblastoma, or medulloepithelioma
* Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that would compromise the patient's ability to tolerate protocol therapy or would likely interfere with the study procedures or results
* Patients receiving any other anticancer or investigational drug therapy, or warfarin
* Patients with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy
* Other: below given criteria are confirmed by the patient history

  * Inability to swallow capsules
  * Malabsorption syndrome or other condition that would interfere with enteral absorption
  * History of congestive heart failure
  * History of ventricular arrhythmia requiring medication
  * Uncontrolled hypocalcemia, hypomagnesemia, hyponatremia or hypokalemia defined as less than the lower limit of normal for the institution despite adequate electrolyte supplementation
  * Clinically important history of liver disease, including viral or other hepatitis or cirrhosis

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11; Primary Completion 2014-06 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amar Gajjar, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (12):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - National Cancer Institute Pediatric Oncology Branch, Bethesda, Maryland
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Robinson GW, Orr BA, Wu G, Gururangan S, Lin T, Qaddoumi I, Packer RJ, Goldman S, Prados MD, Desjardins A, Chintagumpala M, Takebe N, Kaste SC, Rusch M, Allen SJ, Onar-Thomas A, Stewart CF, Fouladi M, Boyett JM, Gilbertson RJ, Curran T, Ellison DW, Gajjar A. Vismodegib Exerts Targeted Efficacy Against Recurrent Sonic Hedgehog-Subgroup Medulloblastoma: Results From Phase II Pediatric Brain Tumor Consortium Studies PBTC-025B and PBTC-032. J Clin Oncol. 2015 Aug 20;33(24):2646-54. doi: 10.1200/JCO.2014.60.1591. Epub 2015 Jul 13. PMID 26169613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was distributed to the sites on 11/22/2010, and received the first IRB approval on 02/02/2011. It was closed to accrual on 03/25/2015. As of the closure date, 42 patients have been pre-screened for Hh pathway activation. Of the 42 patients, 9 patients with Hg pathway activated tumors were registered.
Pre-assignment Details: There were three patients treated at the MTD of GDC-0449 on PBTC-025 who had Hh pathway activated tumors and who met the eligibility criteria for PBTC-032. These three patients were included in the assessment of the primary objectives for PBTC-032.
Groups:
- Hh Pathway Activated: Pediatric patients with recurrent or refractory medulloblastoma with evidence of activation of Hedgehog (Hh) signaling pathway in their tumors.
Period: Overall Study
Arm/Group | Hh Pathway Activated
Started | 12
Completed | 0
Not Completed | 12
Not completed — Progression/Relapse | 11
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Hh Pathway Activated
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] — Age at study enrollment
  years | 10.4 [3.9 to 20.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (CR+PR) Sustained for ≥ 8 Weeks
Description: Objective response is either a complete response or a partial response sustained for 8 weeks in a patient. The objective response rate will be reported separately for patients of each stratum. CR is complete disappearance of all enhancing tumor. PR is >= 50% reduction in tumor size.
Time Frame: Up to 12 months
Measure: Number; unit: participants
Arm/Group | Hh Pathway Activated
Number analyzed (Participants) | 12
participants | 1

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is measured from the date of initial treatment with GDC-0449 until the earliest of progression or death on study. PFS is censored at the last tumor assessment date for patients without disease progression who have not died within 30 days of last exposure to study treatment. Kaplan-Meier method is used to estimate the progression-free survival.
Time Frame: From start of treatment up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Hh Pathway Activated
Number analyzed (Participants) | 12
months | 1.41 [0.69 to 3.68]

3. Primary Outcome: Pharmacokinetics (Plasma) of GDC-0449
Description: plasma GDC-0449 concentration of day 21 in first course
Time Frame: up to 12 month
Population: Patients who have day 21 plasma GDC-0449 concentration data available
Measure: Median (Full Range); unit: uM
Arm/Group | Hh Pathway Activated
Number analyzed (Participants) | 11
uM | 18 [9.5 to 45.3]

4. Secondary Outcome: Duration of Objective Response
Description: The duration of objective response is measured from the initial scan documenting complete or partial response that was subsequently confirmed until the earlier of documented progression or death on study. Duration of objective response is censored at the last tumor assessment date for patients without disease progression who have not died within 30 days of last exposure to study treatment.
Time Frame: From start of treatment up to 2 years
Population: Patient with sustained objective response
Measure: Number; unit: months
Arm/Group | Hh Pathway Activated
Number analyzed (Participants) | 1
months | 2.83

5. Secondary Outcome: Pharmacokinetic Parameters of Vismodegib, CSF Penetration
Description: The estimated median of cerebrospinal fluid (CSF) drug penetration is reported when expressed as an AUC ratio of CSF vismodegib to that of unbound drug in plasma.
Time Frame: up to 12 month
Population: The calculation of drug penetration is based on patients who had the course 1 plasma and CSF drug concentration data
Measure: Median (Full Range); unit: penetration rate
Arm/Group | Hh Pathway Activated
Number analyzed (Participants) | 11
penetration rate | 0.14 [0.07 to 0.28]

ADVERSE EVENTS:
Arm/Group | Hh Pathway Activated
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hh Pathway Activated (N=12)
Lymphocyte count decreased (Investigations) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hh Pathway Activated (N=12)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Blurred vision (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Lip pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6)
Death NOS (General disorders) | 2 (2)
Fatigue (General disorders) | 6 (6)
Gait disturbance (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Lymphocyte count decreased (Investigations) | 2 (4)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Musculoskeletal and connective tissue disorder - Other (Specify, __)[mild cramping in hands.] (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Specify, __)[muscle cramps in calf] (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Specify, __)[Muscle Cramps.] (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other specify[Generalized muscle aches] (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify[Leg muscle cramps] (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify[Muscle spasm/twitching] (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify[MUSCLE SPASMS/TWITCHING] (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify[muscle twitching] (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (4)
Hydrocephalus (Nervous system disorders) | 1 (1)
Movements involuntary (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less